CLINICAL TRIAL: NCT06465498
Title: Investigating ACute HeArt FailuRe Decongestion Guided by Lung UltraSonography (IcarUS) : a Randomized Controlled Trial
Brief Title: Investigating ACute HeArt FailuRe Decongestion Guided by Lung UltraSonography
Acronym: IcarUS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Antonio Leidi (Other)
Collaborators: University Hospital, Geneva (Other)
Responsible Party: Sponsor-Investigator, Antonio Leidi, M.D., Principal Investigator, Attending physician in Internal and Emergency Medicine Services, University Hospital, Geneva
Organization: University Hospital, Geneva (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2024-00268
Record Dates: First submitted 2024-06-13; First posted 2024-06-20 (Actual); Last update posted 2025-03-19 (Actual); Status verified 2024-08

CONDITIONS: Acute Heart Failure
Keywords: Lung ultrasonography; Ultrasound; Point-of-care ultrasonography; Decongestion; Diuretic

STUDY DESIGN:
Intervention Model Description: Multicentric blinded randomized controlled trial (RCT)
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: To reduce the risk of bias several levels of blinding are introduced:
  1. Patients are blinded to their study arm allocation.
  2. Treating physicians are blinded to the patient's study arm (both PE and POCUS arms will benefit from recommendations for decongestive therapy based on a generic congestion score).
  3. Both sonographers and clinical investigators are reciprocally blinded and masked to the patient's study arm and clinical data files.
  4. Outcomes adjudicators are blinded the patient's study arm
  5. The biostatistician is blinded to the patients' study arm
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Lung ultrasonography (LUS) (Experimental): The antero-lateral thorax is examined using an 8-point protocol. Each region is coded positive in presence of ≥3 B-lines simultaneously on a frozen image or in presence of significant pleural effusion (i.e. extending over the costophrenic angle). A 4-level congestion score is defined: absence of congestion (0-1 positive points), mild congestion (2-3 positive points), moderate congestion (4-5 positive points) and severe congestion (6-8 positive points).
  Interventions: Procedure: LUS decongestive strategy
- Physical Examination (PE) (Active Comparator): Congestion is clinically assessed by calculating the Everest score. This score, previously used in clinical trials, is composed of 3 congestion symptoms (i.e. dyspnea, orthopnoea and fatigue) and 3 congestion signs (i.e. jugular vein distension, lung rales, oedema), each graded from 0 to 3. From the total score, a sub-score is derived, ranging from absence of congestion to severe congestion.
  Interventions: Procedure: PE decongestive strategy

INTERVENTIONS:
Procedure: LUS decongestive strategy — LUS results are documented in the electronic case report form (eCRF) and converted into a common score ranging from absence of congestion to severe congestion. This generic congestion score will be communicated to the treating physician by the research personnel, along with a proposal to step-up, maintain, or step-down the decongestive therapy.
  Arms: Lung ultrasonography (LUS)
Procedure: PE decongestive strategy — PE results are documented in the eCRF and converted into a common score ranging from absence of congestion to severe congestion. This generic congestion score will be communicated to the treating physician by the research personnel, along with a proposal to step-up, maintain, or step-down the decongestive therapy.
  Arms: Physical Examination (PE)

SUMMARY:
The goal of this clinical trial is to investigate whether a lung ultrasonography (LUS)-guided decongestion strategy in adults hospitalized for acute heart failure (AHF) can improve patient-centered outcomes.

The main questions it aims to answer are:

* Does this strategy shorten the length of stay and reduce early hospital readmissions?
* Does this strategy improve patients' symptoms and quality of life ?

Researchers will compare LUS to physical examination (PE).

DETAILED DESCRIPTION:
Background: Despite recent medical advances, AHF remains one of the leading causes of hospital admissions and one of the most frequent reasons for readmission. As the main reason for AHF hospitalization is congestion-driven symptoms, the cornerstone of treatment is decongestive therapy. In the absence of specific quantitative measures, however, undertreatment often occurs and is associated with an increased risk of readmission. LUS is highly accurate for detecting extravascular lung water (EVLW). It has shown clinical benefits when used to guide decongestive therapy in chronic heart failure ambulatory patients. However, data for its use in AHF inpatients are currently lacking.

Aim: To investigate the effect of a bedside LUS-guided decongestive therapy in hospitalized AHF adults on patient-centered outcomes, as compared to usual care.

Methodology: This will be a Swiss multicenter, blinded, randomized controlled trial (RCT) aiming to recruit 222 adults hospitalized for congestive acute heart failure (AHF). Study participants will be included within the first 48 hours of their hospital arrival. Patients will be randomized to either a LUS-guided decongestive strategy or a decongestive strategy based on a structured physical examination. The primary outcome will be the number of days spent alive outside the hospital within a 40-day timeframe from study inclusion (DAOH-40). This outcome integrates length of stay, early readmission, emergency room visits, and mortality.

ELIGIBILITY:
Inclusion Criteria:

* ≥ 18 years old
* Planned or actual admission to intermediate care units, general internal medical or cardiology wards
* Diagnosis of congestive AHF on admission chart (primary or secondary diagnosis)
* Raised value of N terminal-pro-brain natriuretic peptide (≥1000 ng/l).

Key Exclusion Criteria:

* Known isolated right heart failure
* Systolic blood pressure <90 mmHg, mean arterial pressure <65 mmHg at the moment of inclusion
* The following conditions mimicking lung cardiogenic oedema on LUS if known at inclusion and documented: Interstitial lung disease, lung cancer or metastasis, acute respiratory distress syndrome, pulmonary contusion
* Known virologically confirmed SARS-CoV-2 pneumonia in the preceding 3 months
* Unwillingness to give consent
* Subjects who are pregnant or breastfeeding
* Hospitalisation for palliative care and probable end-life within 30 days

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 222 (Estimated)
Dates: Start 2024-10-22 (Actual); Primary Completion 2026-08-30 (Estimated); Study Completion 2026-08-30 (Estimated)

PRIMARY OUTCOMES:
DAOH-40 | 40 days from study inclusion
  Number of days spent alive outside the hospital in a 40-day timeframe from study inclusion.
  This outcome ultimately evaluates number of days spent alive and nonhospitalized, simultaneously assessing (re)hospitalization, unplanned emergency visits and mortality

SECONDARY OUTCOMES:
Successful decongestion | 3 working days after randomization
  Proportion of participants obtaining successful decongestion, i.e the absence of signs of volume overload as defined by the Acetazolamide in Decompensated Heart Failure with Volume Overload (ADVOR) congestion score.
Diuretic dose | Uo to 6 working days after randomisation
  Mean daily dose of diuretic therapy during study intervention (in furosemide iv equivalent)
EQ-5D-5L questionary | Up to 90 days after discharge
  Quality of life questionary. EQ-5D-5L index scores range from -0.59 to 1, where 1 is the best possible health state; EQ VAS scores range from 0 to 100, where 100 is the best possible health state.
Readmission and any-cause mortality | Up to 90 days after discharge
  Rate of hospital readmissions and deaths occurring within 90 days of discharge
HF-related hospitalisation | Up to 90 days after discharge
  Rate of HF-related hospitalisation, as defined by the presence of worsening signs and symptoms of HF and an intensification of the diuretic therapy
Length of hospital stay | Through hospitalization, an average of 9 days
  Mean length of hospital stay
Dyspnea | Up to 90 days after discharge
  Dyspnea assessed with a 100-mm Visual Analog Scale (VAS), score ranging from 0 to 100, higher scores mean worse outcome.
Anxiety and depression | Up to 90 days after discharge
  Hospital Anxiety and Depression Scale, two subscales ranging from 0 to 21 points, higher scores mean worse outcome.

OTHER OUTCOMES:
Worsening of renal function | Up to 6 working days after randomisation
  ≥50% rise of serum creatinine from baseline value
Hyponatremia | Up to 6 working days after randomisation
  Rate of severe hyponatremia <120 mmol/l
Hypokaliemia | Up to 6 working days after randomisation
  Rate of severe hypokaliemia <2.5 mmol/l
Sustained hypotension | Up to 6 working days after randomisation
  proportion of patients needing vasopressor/inotropic agents because of sustained hypotension

CONTACTS AND LOCATIONS:
Locations (4):
- Switzerland (4):
  - Geneva University Hospitals, Geneva, Canton of Geneva
  - Inselspital, Universitätspital, Bern, Switzerland
  - Fribourg University Hospital, Fribourg
  - Ospedale Civico, Ente Ospedaliero Cantonale, Lugano

IPD SHARING:
Plan to Share IPD: No